CLINICAL TRIAL: NCT03583892
Title: Use of Preoperative Gabapentin in Patients Undergoing Laparoscopic Cholecystectomy
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Centro Hospitalar do Porto (Other)
Responsible Party: Principal Investigator, Ana Rita Marques Saraiva, Rita Saraiva, Centro Hospitalar do Porto
Other Study IDs: 2017 - 130 (111-DEFI/104-CES)
Record Dates: First submitted 2018-05-10; First posted 2018-07-12 (Actual); Last update posted 2019-08-09 (Actual); Status verified 2019-08

CONDITIONS: Pain, Postoperative
Keywords: Gabapentin, laparoscopic cholecystectomy, postoperative pain
MeSH Terms: conditions — Pain, Postoperative | interventions — Gabapentin

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 1 Day
Oversight: FDA-regulated Drug: Yes

GROUPS / COHORTS (2):
- Group A: In the Group A, a single-dose of 600mg gabapentin was used as part of a multimodal analgesic technique.
  Interventions: Drug: Gabapentin
- Group B: In the group B gabapentin was not administered.

INTERVENTIONS:
Drug: Gabapentin — One of the groups of patients was exposed to preoperative gabapentin. As the pain has a complex involvement of multiple mechanisms, multimodal analgesic techniques utilizing a number of drugs acting on different analgesic mechanisms are being used. In this case, some patients received gabapentin as a part of a multimodal analgesic technique.
  Groups: Group A

SUMMARY:
The multimodal analgesia involves the administration of two or more analgesic agents that exert their effects via different analgesic mechanisms, providing superior analgesia with fewer side effects. This multimodal analgesic regimen includes opioids, nonsteroidal antiinflammatory drugs, cyclooxygenase-2 inhibitors, gabapentinoids, local anesthetics, and peripheral nerve blocks. The aim of this study is to evaluate postoperative analgesic benefit in patients administered with 600mg oral gabapentin as premedication for laparoscopic cholecystectomy under general anesthesia, with respect to postoperative pain scores and total postoperative requirements of morphine and/or tramadol.

DETAILED DESCRIPTION:
Postoperative pain after laparoscopic cholecystectomy is not only nociceptive but also inflammatory, neurogenic and visceral. Therefore, because of involvement of multiple mechanisms, multimodal analgesic techniques utilizing a number of drugs acting on different analgesic mechanisms are being used. The multimodal analgesic mechanisms include opioids, nonsteroidal antiinflammatory drugs, cyclooxygenase-2 inhibitors, gabapentinoids, local anesthetics, and transversus abdominis plane block. Pre-treatment with gabapentin blocks the development of hyperalgesia and tactile allodynia for up to two days. The aim of this study is to evaluate postoperative analgesic benefit in patients administered with 600mg oral gabapentin as premedication for laparoscopic cholecystectomy under general anesthesia, with respect to postoperative pain scores and total postoperative requirements of morphine and/or tramadol. In the preoperative period, consent is requested for patients who meet the inclusion criteria of the study. At this time it is verified whether gabapentin has been prescribed by the attending physician or not. If enrolled, the patient is allocated to the gabapentin group (Group A) or to the non-gabapentin group (Group B), according to his/her prescription.

All patients are monitored for electrocardiogram, pulse oximetry, noninvasive blood pressure, capnography, bispectral index (BIS®), and neuromuscular transmission with Train-of-Four (TOF®) during intraoperative period. Anesthesia is induced with intravenous fentanyl 1 to 3 µg/kg and propofol 1 to 3 mg/Kg. Muscle relaxation is achieved with rocuronium 0.5 to 1,2 mg/Kg and orotracheal intubation is performed when TOF count had reached 0. Anesthesia is maintained with Desflurane and Air/Oxygen, titrated to maintain the BIS value between 40-60. Muscle relaxation is maintained with rocuronium bolus (10mg), when more than two responses are detected in TOF stimulation. The lungs are mechanically ventilated and adjusted to maintain end-tidal carbon dioxide between 35 and 45 mmHg. All patients are given a continuous infusion of polyelectrolyte solution. At the end of surgery, neuromuscular block is antagonized with standard doses of sugammadex (2mg/Kg, if TOF≥2; 4mg/Kg if TOF=0 and Post-Tetanic-Count (PTC) ≥2; 16mg/Kg, if TOF=0 and PTC<2). The endotracheal tube is removed when the TOF ratio is > 90% and BIS > 80, with the patient being conscious, with adequate spontaneous ventilation and responded to verbal commands. Perioperative analgesia is provided with intravenous paracetamol 1g (administrated after anesthetic induction), parecoxib 40mg (administrated after anesthetic induction) and local anesthetic infiltration of trocar insertion sites with ropivacaine 0.5%. When gabapentin is preoperative given, the usual doses is 600mg. Postoperative nausea and vomiting prophylaxis are assured with intravenous dexamethasone 4mg after the induction, and intravenous ondansetron 4mg at the end of the surgery.

At the postanesthesia care unit (PACU), the pain is assessed using a numeric pain rating scale at the arrival (0h) and then at 1, 6, 12, 24h, both at rest and at movement (with a maximum of 30minute variation at each evaluation time). The investigators will also consult the nursing evaluation of pain scores (assessment of pain scores at intervals of 4hours). Patients with sedation score of at least 4 are considered sedated. The occurrence of postoperative complications is also recorded. At any time, if analgesia is inadequate, the anesthesia resident will provide intravenous bolus of morphine (0.05-0.1 mg/Kg) and stop if patient has respiratory depression (defined as respiratory rate<10 per minute or Blood Oxygen Saturation (SpO2)<90% on air) or is sedated. Droperidol 0.625mg will be given intravenously if patient had persistent nausea or had two or more episodes of retching or vomiting. Total consumption of morphine during the stay at the PACU is recorded. - Post-operative analgesia is usually provided with intravenous paracetamol 1g 8/8h and intravenous parecoxib 40mg 12/12h. If the patient still complained of pain, then rescue analgesia will be given with intravenous tramadol 100mg, maximum 8/8h. Besides that, nausea and vomiting prophylaxis are assured with intravenous ondansetron 4mg 8/8h. Total consumption of tramadol during the stay at the ward is recorded.

ELIGIBILITY:
Inclusion Criteria:

* Patients belonging to American Society of Anesthesiologists physical status I and II;
* Patients undergoing elective laparoscopic cholecystectomy, under general anesthesia;
* Age between 18 and 75 years;
* Patients hemodynamically stable.

Exclusion Criteria:

* Patients with an age older than 75 years or younger than 18 years;
* Uncontrolled concomitant medical diseases (hypertension, bronchial asthma, diabetes mellitus);
* Patients with history of chronic pain conditions;
* Impaired kidney or liver function;
* History of drug or alcohol abuse;
* Occurrence of surgical complications that force a change in the established surgical approach;
* Administration of analgesics within 24 hours of scheduled surgery;
* Patients already on gabapentin or other anticonvulsants.

Ages: 18 Years to 75 Years | Sex: All
Age Groups: Adult, Older Adult
Study Population: Patients undergoing elective laparoscopic cholecystectomy in the "Centro Hospitalar do Porto".
Sampling Method: Non-Probability Sample
Enrollment: 60 (Estimated)
Dates: Start 2018-07-01 (Actual); Primary Completion 2020-07 (Estimated); Study Completion 2020-07 (Estimated)

PRIMARY OUTCOMES:
Evaluate postoperative analgesic benefit in patients administered with 600mg oral gabapentin as premedication for laparoscopic cholecystectomy under general anesthesia, with respect to postoperative pain scores, in five different time points. | Postoperative pain is assessed at the arrival (0h) and then at 1, 6, 12, 24h, both at rest and at movement (with a maximum of 30minute variation at each evaluation time).
  Postoperative pain will be evaluated using the Numeric Pain Rating Scale (with minimum and maximum scores varying from 0 to 10, respectively, where 0 means no pain and the value 10 represents the worst imaginable pain). Investigators will also consult the nursing evaluation of pain scores (assessment of pain scores at intervals of 4hours). Higher values represent a worse outcome.

SECONDARY OUTCOMES:
evaluate postoperative analgesic benefit in patients administered with 600mg oral gabapentin as premedication for laparoscopic cholecystectomy under general anesthesia, with respect to total postoperative requirements of morphine and/or tramadol. | Total requirements of morphine and/or tramadol will be recorded during the first 24h of postoperative.
  Total postoperative consumption of morphine and/or tramadol will be recorded in milligrams.

OTHER OUTCOMES:
The presence of postoperative complications, as somnolence, postoperative nausea and vomiting, dizziness, sedation and pruritus. | The first 24h of postoperative.

CONTACTS AND LOCATIONS:
Overall Officials: Rita Saraiva, MD, Principal Investigator — Centro Hospitalar do Porto, Serviço de Anestesiologia
Locations (1):
- Centro Hospitalar do Porto, Porto, Portugal

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Result] Srivastava U, Kumar A, Saxena S, Mishra AR, Saraswat N, Mishra S. Effect of preoperative gabapentin on postoperative pain and tramadol consumption after minilap open cholecystectomy: a randomized double-blind, placebo-controlled trial. Eur J Anaesthesiol. 2010 Apr;27(4):331-5. doi: 10.1097/EJA.0b013e328334de85. PMID 19935070